CLINICAL TRIAL: NCT06631430
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 3810477 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Different Doses of BI 3810477 Are Tolerated by Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1530-0001; 2024-513419-28-00 (Registry Identifier: CTIS); U1111-1306-7752 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A: BI 3810477 formulation A dose group 1 (Experimental): single dose group 1
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 2 (Experimental): single dose group 2
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 3 (Experimental): single dose group 3
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 4 (Experimental): single dose group 4
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 5 (Experimental): single dose group 5
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 6 (Experimental): single dose group 6
  Interventions: Drug: BI 3810477
- Part A: BI 3810477 formulation A dose group 7 (Experimental): single dose group 7
  Interventions: Drug: BI 3810477
- Part B: BI 3810477 formulation B dose group 1 (Experimental): single dose group 1
  Interventions: Drug: BI 3810477
- Part B: BI 3810477 formulation B dose group 2 (Experimental): single dose group 2
  Interventions: Drug: BI 3810477
- Part B: BI 3810477 formulation B dose group 3 (Experimental): single dose group 3
  Interventions: Drug: BI 3810477
- Part A and Part B_Placebo (Placebo Comparator): single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 3810477 — BI 3810477 formulation A
  Arms: Part A: BI 3810477 formulation A dose group 1; Part A: BI 3810477 formulation A dose group 2; Part A: BI 3810477 formulation A dose group 3; Part A: BI 3810477 formulation A dose group 4; Part A: BI 3810477 formulation A dose group 5; Part A: BI 3810477 formulation A dose group 6; Part A: BI 3810477 formulation A dose group 7
Drug: BI 3810477 — BI 3810477 formulation B
  Arms: Part B: BI 3810477 formulation B dose group 1; Part B: BI 3810477 formulation B dose group 2; Part B: BI 3810477 formulation B dose group 3
Drug: Placebo — Placebo
  Arms: Part A and Part B_Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 3810477 in healthy male subjects.

ELIGIBILITY:
Inclusion criteria

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 60 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
4. Signed and dated written informed consent in accordance with international conference on harmonization-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial
5. Male subjects who are willing to use condoms to prevent unintended exposure of their partner (both, male and female) from time point of administration of trial medication until completion of the trial

Exclusion criteria

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 100 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Further exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | Up to Day 85

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 85
Maximum measured concentration of the analyte in plasma (Cmax) | Up to Day 85

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com